CLINICAL TRIAL: NCT02382705
Title: Clinical Impact of Longer Battery Life on Small Bowel Capsule Endoscopy: a Prospective Observational Study
Brief Title: SB3 Battery Life Observational Study
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Robert Enns, Clinical Professor, University of British Columbia
Other Study IDs: H14-03253
Record Dates: First submitted 2015-03-03; First posted 2015-03-09 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2018-12

CONDITIONS: Capsule Endoscopy
Keywords: capsule endoscopy; battery life; completion rate; diagnostic yield

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Capsule endoscopy (CE) is a non-invasive means of visualizing the small bowel. Common indications for CE include obscure gastrointestinal (GI) bleeding, inflammatory bowel disease like crohn's disease or ulcerative colitis, celiac disease, and polyposis syndrome.

While CE has high diagnostic value for small bowel lesions, a significant limitation of this technology is the finite battery life which results in incomplete examination of the small bowel approximately 16.5% of the time. Numerous attempts of using pharmacological (e.g. prokinetics, purgatives) as well as non-pharmacological measures (e.g. real-time viewer, chewing gum) to improve completion rates, defined by entry of CE into the cecum, led to mixed results. Currently routine use of prokinetics (agents that speeds up gut motility) is not recommended.

This study aims to determine whether longer battery of the newer generation capsule endoscopy system improves study completion rate and diagnostic yield.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 19 or greater who are referred for small bowel capsule endoscopy
* Willing and able to provide written informed consent

Exclusion Criteria:

* Unwillingness or inability to swallow pill
* Known or suspected obstruction or bowel stricture
* Endoscopic placement of capsule camera
* Concomitant enrollment in a prospective study in the treatment arm receiving prokinetics for the purpose of enhancing bowel motility. (i.e. control arm not receiving any motility-enhancing agent can be included)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing small bowel capsule endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Enns, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- PillCam SB3EX: All participants in the study used the PillCam SB3EX for their capsule endoscopy
Period: Overall Study
Arm/Group | PillCam SB3EX
Started | 57
Completed | 33
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | PillCam SB3EX
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 57

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate (Rate at Which Small Bowel is Completely Examined)
Description: rate at which small bowel is completely examined (capsule endoscopy enters cecum)
Time Frame: 0.1 - 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | PillCam SB3EX
Number analyzed (Participants) | 57
Participants | 57

2. Secondary Outcome: Diagnostic Yield
Description: rate at which a pathological finding is identified on capsule endoscopy
Time Frame: 0.1 - 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | PillCam SB3EX
Number analyzed (Participants) | 57
Participants | 20

3. Secondary Outcome: Gastric Transit Time
Description: time it takes for capsule camera to traverse the stomach
Time Frame: 0.1 - 12 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PillCam SB3EX
Number analyzed (Participants) | 33
minutes | 37.6 (92.1)

4. Secondary Outcome: Small Bowel Transit Time
Description: times it takes for capsule camera to traverse the entire small bowel.
Time Frame: 0.1 - 12 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PillCam SB3EX
Number analyzed (Participants) | 33
minutes | 232.1 (98.3)

ADVERSE EVENTS:
Groups:
- PillCam SB3EX: Patients who were eligible to participate in the study were recruited and enrolled. Enrolled participants were given instructions for capsule endoscopy as per standard of practice at our institution. External sensors and data recorder for use with the PillCam capsule were placed. Patients swallowed the capsule. All capsule endoscopy were allowed to run/record until the recording terminates due to battery outage (usually after 12 h) or passage of CE out of the gastrointestinal tract, as indicated by cessation of flashing light on the recorder. External sensors and data recorder were removed at the end of the recording and patients returned the equipment to the institution the next day.
Arm/Group | PillCam SB3EX
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No